CLINICAL TRIAL: NCT02550730
Title: Birth Sisters Best Beginnings Evaluation
Brief Title: Best Beginnings for Babies Birth Sister Program Evaluation
Acronym: BBB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Julie Mottl-Santiago, Midwife and Assistant Professor, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-33788
Record Dates: First submitted 2015-06-23; First posted 2015-09-15 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Birth Sisters (Experimental): Half of the women who agree to participate in the evaluation will be randomized to the Birth Sisters Best beginnings for Babies Program, which includes community doula support and consultation with Medical Legal Partnership when indicated.
  Interventions: Behavioral: Birth Sisters Best Beginnings for Babies
- Routine care (Active Comparator): Half of the women who agree to participate in the evaluation will be randomized to the usual maternity care group
  Interventions: Other: Usual maternity care

INTERVENTIONS:
Behavioral: Birth Sisters Best Beginnings for Babies — Birth Sisters Best Beginnings for Babies support during Pregnancy, Labor and Delivery and six weeks postpartum. Participants assigned to the Birth Sister group receive community doula services with consultation from the Medical Legal Partnership when indicated beginning at 24 weeks. Participants receive up to 8 two-hour prenatal home visits; continuous support through labor and birth, and up to 4 two-hour postpartum home visits through 6-8 weeks postpartum.
  Arms: Birth Sisters
Other: Usual maternity care — Usual prenatal, intrapartum and postpartum maternity care
  Arms: Routine care

SUMMARY:
Peer support during labor, birth and the perinatal period (also known as "doula" support) has been shown in some studies to reduce cesarean rates, postpartum depression and increase breastfeeding rates. The purpose of this program evaluation is to prospectively assess the clinical and cost outcomes of Boston Medical Center's Birth Sister doula program, one of the few established, hospital-based programs in the United States. To enhance the capability of the Birth Sisters Program to impact social determinants of perinatal health in a low-income population, the program evaluation will include the addition of Medical Legal Partnership for Children's (MLP) training and referral services. This program will be described as the Birth Sisters Best Beginnings services (BBB). The evaluation will compare the effects of BBB compared with no Birth Sister support for women receiving maternity care at Boston Medical Center. Eligible women will be randomly assigned either BBB services or usual care. All women will be consented and interviewed in the mid-second trimester of pregnancy and interviewed again at 6-8 weeks postpartum. Women randomized to the BBB will be offered 8 prenatal Birth Sister visits in the home or at Boston Medical Center starting at 6 months of pregnancy, continuous support through labor and birth, and up to 4 postpartum Birth Sister visits in the home or at Boston Medical Center. The usual care group will receive no birth sister support but does have access to standard interdisciplinary maternity care services. The primary outcomes will be reduction in cesarean rate. Secondary outcomes will include cost, labor interventions, infant outcomes, satisfaction with care and psychosocial outcomes, including depression, social functioning and self-efficacy.

DETAILED DESCRIPTION:
Racial and income disparities in maternal and perinatal outcomes in the United States are large and persistent. Maternal and infant morbidity and mortality alike are 2-3 times higher in the black population than in the white population. Poor women in general are more likely to have babies born prematurely or with low birth weight compared with women from a higher socio economic strata. Infants born either too early or too small are at risk for a lifetime of disabilities, perpetuating the cycle of poverty and poor health. Low-income and minority populations are also less likely to breastfeed, putting children and mothers at higher risk for a variety of health problems, including obesity, diabetes, and some cancers.

In addition to income and racial disparities, the nation as a whole struggles with inferior maternity care outcomes when compared with other developed countries. This is true despite considerably higher rates of maternity care expenditures. The unnecessarily high rate of cesarean birth is one factor that contributes to both high cost and poor outcomes. The Society of Maternal and Fetal Medicine and the American Congress of Obstetricians and Gynecologists have both called for innovations and strategies to reduce the high rate of cesarean birth.

Community "doulas", or peer support during pregnancy, labor and birth, is one intervention that may both improve outcomes for low-income populations and lower the cost of maternity care. A culturally competent peer who provides caring support during a crucial life transition may lower stress and improve engagement in healthcare, therefore improving health status during pregnancy and lowering the need for costly medical care. Low income and minority women are more likely to desire a doula during labor and less likely to have access to their services.

The Birth Sisters Program One of the few hospital-based community doula programs in the country, Boston Medical Center's Birth Sisters Program has provided multicultural doula support to childbearing women since 1999. The approximately 20 per diem Birth Sisters together speak over 10 languages. Birth Sisters are recruited from the communities served by the BMC maternity service and provide peer support throughout the perinatal period. Prenatal home visits focus on creating a relationship, identifying psychosocial needs and providing childbirth and breastfeeding education. The Birth Sister also assesses whether the woman is lacking in essential resources such as housing, food and baby care items. She then refers her client to social service agencies and helps her navigate those services as needed. During labor, the Birth Sister offers physical and emotional comfort measures, advocacy for the mother, and help with the first breastfeeding. Postpartum home visits provide assistance in the transition to motherhood, help around the house so that the mother can rest, education on breastfeeding, parenting and infant care, and connections to needed medical and social services.

The Birth Sisters Program does not have resources to serve all women who would like a Birth Sister. investigators are currently able to meet approximately 20 percent of the demand. Prenatal providers have traditionally been the primary referral source for the program, with some providers referring often and others rarely referring. This has created inequities in whether women have a chance to receive a Birth Sister. investigators are now changing the referral process to systematically screen all potentially eligible women and allow eligible women to self-refer to the Birth Sister pool. A limited number of Birth Sister assignments are made from this pool each month. Women are informed about the Birth Sister pool through flyers placed in the obstetrical ultrasound unit and, if they would like to be in the pool, they fill out a form with their contact information and place it in the "Birth Sister pool" box. Due to the budget limitations, investigators restrict referrals to women who benefit most, including first time mothers with public insurance.

Because investigators only have resources to serve a small portion of women who want a Birth Sister, investigators have designed an evaluation to provide rigorous evidence about the health and economic outcomes of our program. Prospective, high-quality data is needed to inform policy questions about the benefits of billable community doulas for Medicaid recipients. This is our justification for randomization in a study testing a standard care program.

Purpose The primary objective of the proposed project is to determine the effectiveness of the Birth Sisters Program, in reducing cesarean birth rates and cost of care in a safety net population. The associated objectives are, by the end of the project, to demonstrate significant reductions in: depressive symptoms, low birth weight and preterm birth; and significant increases in breastfeeding rates in women accessing enhanced Birth Sisters as compared to women who are not supported by Birth Sisters. Effective interventions must be sustainable. Cost of care analyses will evaluate whether the incremental costs of the Birth Sisters Program services are justified by the savings brought about by lower rates of labor complications, cesarean sections, emergency room visits and NICU days.

Of note, to improve the ability of the Birth Sisters to address social determinants of health, this evaluation will add training and consultations for Birth Sisters and their clients by Medical Legal Partnership (MLP). MLP is a team of legal experts who integrate legal assistance into the medical setting as a vital component of patient care to ensure that low-income patients are able to meet legal needs that impact on health. They will provide trainings for Birth Sisters on key legal issues, such as housing and benefits. They will also be available for consultation when the mother requires additional resources and information.

Investigators hypothesize that women receiving the BBB intervention will:

1. exhibit lower rates of cesarean sections, low birth weight and preterm birth, and neonatal intensive care unit days; and
2. exhibit the highest rates of breastfeeding initiation, exclusivity, and continuation;
3. experience reductions in depressive symptoms;
4. incur lower health care costs than incremental program costs, providing evidence for long-term sustainability.

ELIGIBILITY:
Inclusion criteria:

* Being a pregnant Woman 16 to 24 gestational age
* First Time Mother
* Singleton
* Public insurance
* No known fetal anomaly

Exclusion criteria

* < 18 years of age
* high risk pregnancy defined by care in the high-risk prenatal clinic

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 411 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Rates of cesarean sections | at delivery
  total cesareans/total births as assessed by medical record abstraction

SECONDARY OUTCOMES:
Rates of preterm birth | at delivery
  total preterm births/total births as assessed by medical record abstraction

OTHER OUTCOMES:
Low birth weight, | at delivery
  total births<2500g/total births as assessed by medical record abstraction
Rates of breastfeeding initiation | 8 weeks postpartum
  Number of mothers initiating breastfeeding/total # mothers by medical record abstraction
Reductions in depressive symptoms | 8 weeks postpartum
  Number of mothers with depression scale scores>9/total # mothers
Lower health care costs than incremental program costs | 8 weeks postpartum
  medical center costs reported through hospital accounting system
Rates of breastfeeding continuation | 8 weeks postpartum
  percent of participants breastfeeding at 8 weeks postpartum by interview
Rates of breastfeeding exclusivity | 8 weeks postpartum
  percent of participants exclusively breastfeeding at 8 weeks pp by interview

CONTACTS AND LOCATIONS:
Overall Officials: Julie Mottl-Santiago, MPH, CNM, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mottl-Santiago J, Dukhovny D, Cabral H, Rodrigues D, Spencer L, Valle EA, Feinberg E. Effectiveness of an Enhanced Community Doula Intervention in a Safety Net Setting: A Randomized Controlled Trial. Health Equity. 2023 Sep 7;7(1):466-476. doi: 10.1089/heq.2022.0200. eCollection 2023. PMID 37731785